CLINICAL TRIAL: NCT06676202
Title: The Effect of Progressive Relaxation Exercises on Anxiety Levels in Patients Undergoing Total Knee Replacement Surgery: a Randomized Controlled Trial
Brief Title: Progressive Relaxation Exercises on Anxiety Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Meryem FIRAT, Erzincan University, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ramazan_YENİ_YL_TEZ
Record Dates: First submitted 2024-10-16; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Exercises Therapy; Total Knee Replacement Surgery
Keywords: Anxiety; Exercises; Total Knee Replacement Surgery
MeSH Terms: conditions — Anxiety Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: The sample will not be selected from the universe and all patients who meet the inclusion criteria will constitute the sample. The minimum sample size of the study was determined by performing power analysis with the G-power 3.1.9.4 program. In the calculation made according to the two-way independent samples t-test, the effect size was taken as 0.80, with a margin of error of 0.05 and a power of 90%, the total sample number was calculated as 60 (Cohen, 1998). Considering the losses within the scope of the study, 66 patients who meet the inclusion criteria will be randomly divided into the experimental group (33 patients) and the control group (33). Finally, in order to minimize the risk of contamination, the first 33 patients who meet the inclusion criteria after being admitted to the clinic will constitute the control group, and the following 33 patients will constitute the experimental group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): - The patient will be given progressive relaxation exercises at the 12th, 24th, and 48th hours after the surgery. Before the application, information will be obtained about whether the patient has any complications and patients who develop complications due to the surgery will be excluded from the research group. As a result of the screening of progressive relaxation exercise studies in the literature, no standard duration and frequency information was found regarding the effectiveness of progressive relaxation exercise (Haut et al, 2018). In the literature review, it is seen that the total number of sessions varies as well as different applications such as being applied at the 6th, 12th, 24th hours after surgery or on the 2nd day after surgery (Tanrıverdi, 2021). In addition, studies conducted to reduce anxiety, pain, and stress after surgery may vary according to the length of hospitalization (Sertbaş and Bahar, 2004). Based on this information, it was learned that the approximate h
  Interventions: Behavioral: Progressive Relaxation Exercises
- Control Group (No Intervention): * After the 33 patients admitted to the clinic, the "Patient Introduction Form" and "Beck Anxiety Scale" will be filled out after information and consent.
  * After the total knee replacement surgery, 50 hours will be waited and then the "Patient Introduction Form" and "Beck Anxiety Scale" will be filled out again.
  * Progressive relaxation exercises will not be applied to the control group patients, but the pre-test and post-test data will be applied in the same time periods as the experimental group.
  * Pre-test application 1 day before the surgery (Since the patient may be too tense just before the surgery, 1 day before was preferred. Patients who are taken to surgery on the same day due to an emergency will be excluded from the research group.)
  * Post-test application 50 hours after the surgery and later (Relaxation exercises will be applied to the experimental group at 12-24 and 48 hours. The 48th hour, when the exercise ends, will not be preferred for the post-test, the patient

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises — It combines the contraction and relaxation of large muscle groups such as the face, arms, legs, neck and back with deep breathing exercises. Before applying progressive relaxation exercises, the environment should be quiet, dimly lit, a comfortable chair or armchair should be sat or lying down, and clothing should be loose and comfortable, and it is recommended to apply it one hour after eating. In the application of progressive relaxation exercises, it is first asked to breathe regularly. After our breathing rhythm is regulated, the hands, arm muscles, shoulder and neck muscles, chest, abdominal and hip muscles, legs, feet and facial muscles are contracted with a 5-7 second breathing exercise and relaxed during exhalation. This is repeated with 4-5 breathing exercises for each muscle and the exercise is ended when the eyelids are opened.
  Arms: Experimental group

SUMMARY:
The research will be conducted to determine the effect of progressive relaxation exercises on the anxiety level of patients who have had total knee replacement surgery.

DETAILED DESCRIPTION:
The sample will not be selected from the universe and all patients who meet the inclusion criteria will constitute the sample. The minimum sample size of the study was determined by performing power analysis with the G-power 3.1.9.4 program. In the calculation made according to the two-way independent samples t-test, the effect size was taken as 0.80, with a margin of error of 0.05 and a power of 90%, the total sample number was calculated as 60 (Cohen, 1998). Considering the losses within the scope of the study, 66 patients who meet the inclusion criteria will be randomly divided into the experimental group (33 patients) and the control group (33). Finally, in order to minimize the risk of contamination, the first 33 patients who meet the inclusion criteria after being admitted to the clinic will constitute the control group, and the following 33 patients will constitute the experimental group.

Data will be collected using the 'Patient Identification Form' and the 'Beck Anxiety Scale'.

Progressive relaxation exercises were first applied by Dr. It is a technique of voluntary muscle contraction and relaxation developed by Edmund Jacobson in the 1920s. The main purpose of progressive relaxation exercises is for patients to understand the difference between muscle relaxation and tension and to be able to relax on their own. It combines the contraction and relaxation of large muscle groups such as the face, arms, legs, neck and back with deep breathing exercises. Before applying progressive relaxation exercises, the environment should be quiet, dimly lit, in a comfortable chair or armchair, sitting or lying down, and clothing should be loose and comfortable, and it is recommended to apply it one hour after eating. In the application of progressive relaxation exercises, it is first asked to breathe regularly. After our breathing rhythm is regulated, the hands, arm muscles, shoulder and neck muscles, chest, abdominal and hip muscles, legs, feet and facial muscles are contracted with a 5-7 second breathing exercise and relaxed during exhalation. This is repeated with 4-5 breathing exercises for each muscle and the exercise is ended when the eyelids are opened.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old and above
* Speaking and understanding Turkish
* Having total knee replacement surgery
* Staying in the ward for approximately 96 hours after surgery
* Volunteering to participate in the study
* Not having a psychiatric diagnosis

Exclusion Criteria:

* Being under 18 years old
* Having speech and comprehension problems
* Not having total knee replacement surgery
* Early discharge after surgery
* Having complications after surgery
* Not volunteering to participate in the study
* Having a psychiatric diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Progressive relaxation exercises do not affect the anxiety level in patients who underwent total knee arthroplasty. | at the 12th, 24th and 48th hours after surgery
  In order to assess the anxiety level of the patients, the Beck Anxiety Scale will be administered at the 12th, 24th and 48th hours after surgery.
The anxiety level decreases after progressive relaxation exercises in patients who have undergone total knee arthroplasty. | at the 12th, 24th and 48th hours after surgery
  In order to assess the anxiety level of the patients, the Beck Anxiety Scale will be administered at the 12th, 24th and 48th hours after surgery.
The anxiety level increases after progressive relaxation exercises in patients who have undergone total knee arthroplasty. | at the 12th, 24th and 48th hours after surgery
  In order to assess the anxiety level of the patients, the Beck Anxiety Scale will be administered at the 12th, 24th and 48th hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yildirim Universty, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No